CLINICAL TRIAL: NCT07150754
Title: Heart Failure Pharmacological Treatments and Falls in Older Adults: A Disproportionality Analysis of the WHO Pharmacovigilance Database
Brief Title: Cardiological Drug Classes And Falls in Older Adults
Status: Completed | Type: Observational
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: PHARMACOGERIA092025
Record Dates: First submitted 2025-08-25; First posted 2025-09-02 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Heart Failure; Fall
Keywords: Heart failure; Falls; Pharmacological treatments
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Heart failure pharmacological treatments — Identify a positive signal for fall with one or more of the recommended pharmacological treatments for heart failure

SUMMARY:
Heat failure is a fast gowing health issue with a rising incidence in older adults. Recommendations have recently been published to treat heart failure, but most clinical trials leading to these recommendations tended to exclude older adults.

Older adults are at higher risk of falls and severe consequences of falls. All heart failure treatments are at risk of causing a fall through different mechanisms.

Based on the World Health Organization global database, the main objective of this study is to investigate the association between heart failure pharmacological treatments and the report of a fall in the database.

A disproportionality analysis will be performed. It will aim to assess whether some classes of heart failure drugs, and within these classes some individual drugs, are associated with a report of a fall.

A sensibilty analysis will also be performed. It will aim to examine the association between takien a heart failure pharmacological treatment, with a heat failure indication and/or a loop diuretic, and the report of a fall.

ELIGIBILITY:
Inclusion Criteria:

* Age 65 years of older

Exclusion Criteria:

-

Min Age: 65 Years | Sex: All
Age Groups: Older Adult
Study Population: Patients aged 65 years and over who presented fall with one or more recommended heart failure drugs
Sampling Method: Non-Probability Sample
Enrollment: 100000 (Actual)
Dates: Start 2024-11-02 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
Report of a fall with a recommended pharmacological treatment for heart failure | 02/11/2024

SECONDARY OUTCOMES:
Sensibility analysis | 02/11/2024
  Reports of falls with one or more of the respective drug classes that also had either "furosemide" prescription and/or "heart failure" as indication

CONTACTS AND LOCATIONS:
Locations (1):
- Caen University Hospital, Department of Pharmacology, Caen, Normandy, France